CLINICAL TRIAL: NCT03579979
Title: To Evaluate the Safety and Efficacy of Near-infarred Fluorescence Molecular Imaging in the Prospective, Multi-center and Self-controlled Clinical Trial of Sentinel Lymph Node Biopsy in Breast Cancer Surgery
Brief Title: Sentinel Lymph Node Biopsy in Breast Cancer Surgery Using ICG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Beijing Digital Precesion Medicine Company (Unknown); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Friendship Hospital (Other); Tangshan People's Hospital (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Chongwei Chi, Ph.D, Associate Professor, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-DPM-02
Record Dates: First submitted 2018-06-08; First posted 2018-07-09 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Sentinel Lymph Node; Breast Cancer
Keywords: Near-infrared fluorescence; Image guided surgery; Sentinel lymph node biopsy; Indocyanine green; Methylene blue
MeSH Terms: conditions — Breast Neoplasms | interventions — Methylene Blue; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self control (Experimental): During the operation, with the fluorescent molecular imaging instrument, the imaging agent (indocyanine green) is illuminated by the probe distance to the tissue surface 10-30cm, and is excited to produce the near infrared fluorescence of the specific wavelength (the human eye is not visible). The system uses a photoelectric coupler to collect the light of the specific spectrum, and the image is collected by the method of correction. The operation was performed to achieve real-time display of lesions.
  The injection points were selected subcutaneously around the areola or the periphery of the tumor. 1% methylene blue 0.5ml was injected at each point, with a total of 2-3 points. Within 5 minutes, 2.5mg/ml ICG 0.5ml was injected at each point, with a total of 2-3 points.
  Interventions: Drug: Methylene Blue; Drug: Indocyanine Green

INTERVENTIONS:
Drug: Methylene Blue — Subcutaneous injection of injection point at the periphery of the areola or tumor, injecting 1% methylene blue 0.5ml at each point, a total of 2-3 points.
  Other Names: MB
Drug: Indocyanine Green — Within 5 minutes after MB injection, 2.5mg/ml ICG 0.5ml was injected at each point, a total of 2-3 points. Methylene blue and ICG injection points do not coincide
  Other Names: ICG

SUMMARY:
This clinical trial is a prospective, multicenter, self-controlled clinical study. In order to meet the requirements of this plan, 130 breast cancer patients need the sentinel lymph node biopsy with novel near-infarred fluorescence imaging system produced by Beijing digital precision medical technology co., LTD. The fluorescence molecular imaging of indocyanine green (ICG) on imaging detection and the control group, routine medical using methylene blue test .The safety and efficacy of fluorescence and staining in sentinel lymph node biopsy of breast cancer were compared.

DETAILED DESCRIPTION:
This trial was a prospective, multicenter, and self controlled clinical trial. The subjects who were in line with this scheme were detected by fluorimetry and staining, and the primary effectiveness evaluation index, secondary effectiveness evaluation index and safety evaluation index were established during the operation. Record evaluation. At present, in the clinic for sentinel lymph node biopsy of breast cancer, routine medical treatment is a blue staining method. A large number of clinical data show that the number of blue staining methods was 1-2.4, and the number of fluorescence detection is 2-3.7. Therefore, choosing a self controlled clinical trial can increase the number of sentinel lymph node detection.

ELIGIBILITY:
Inclusion Criteria:

1. the age of 18-75 years, female patients;
2. the diagnosis of breast cancer by biopsy;
3. participants voluntarily participated in the clinical trial and signed informed consent.

Exclusion Criteria:

1. had received SLNB or axillary surgery;
2. breast area radiotherapy or neoadjuvant chemotherapy has been accepted.
3. clinical hints of axillary lymph node metastasis;
4. discovery of distant metastasis;
5. inflammatory breast cancer;
6. women in pregnancy;
7. people with iodine allergy;
8. the serum creatinine was > 1.5 times as high as the upper limit of the normal value.
9. to participate in clinical trials of other devices or drugs within one month;
10. the researchers consider it inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node detection number | 1 year
  Participants will be followed for the duration of hospital stay, an expected average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] He K, Chi C, Kou D, Huang W, Wu J, Wang Y, He L, Ye J, Mao Y, Zhang GJ, Wang J, Tian J. Comparison between the indocyanine green fluorescence and blue dye methods for sentinel lymph node biopsy using novel fluorescence image-guided resection equipment in different types of hospitals. Transl Res. 2016 Dec;178:74-80. doi: 10.1016/j.trsl.2016.07.010. Epub 2016 Jul 18. PMID 27497181
- [Result] Chi C, Ye J, Ding H, He D, Huang W, Zhang GJ, Tian J. Use of indocyanine green for detecting the sentinel lymph node in breast cancer patients: from preclinical evaluation to clinical validation. PLoS One. 2013 Dec 16;8(12):e83927. doi: 10.1371/journal.pone.0083927. eCollection 2013. PMID 24358319